CLINICAL TRIAL: NCT00158691
Title: A Randomized Phase III Study Comparing Intravenous Versus Subcutaneous Administration of Amifostine in Prevention of Xerostomia for Patients Receiving Radiotherapy for Head and Neck Carcinomas
Brief Title: Intravenous Versus Subcutaneous Amifostine in Prevention of Xerostomia After RT for Head and Neck Carcinomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2000-02
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck cancer; Radiotherapy; Xerostomia; Randomized trial
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia | interventions — Amifostine

INTERVENTIONS:
Drug: Ethyol

SUMMARY:
Prospective randomized study in order to compare intravenous versus subcutaneous administration of amifostine in patients receiving radiotherapy for head and neck cancer. Salivary flow will be evaluated during few years after the treatment by a clinical evaluation, the measure of the weight of saliva and a patient benefit questionnaire cotation.

DETAILED DESCRIPTION:
Prospective randomized study in order to compare intravenous (IV) versus subcutaneous (SC) administration of amifostine in patients receiving radiotherapy for head and neck cancer. IV administration of amifostine is 200 mg/m2/day in a short 3-min infusion 15 to 30 min before each fraction of radiotherapy. SC administration is 500mg/day in two slow 1.25 ml injections at two different sites 20 to 60 min before each radiotherapy fraction. Procedure requires antiemetic treatment and blood pressure monitoring in both arms.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed squamous cell head and neck cancer
* inclusion of at least 75% of both parotid glands within radiation fields that would receive at least 40 Gy
* Neutrophils ≥ 2000 / mm, Platelets ≥ 100,000 / mm3, Creatinine < 130 / mmol.L-1, Transaminase ≤ 3 x upper limit

Exclusion Criteria:

* Distant metastases
* Prophylactic use of pilocarpine
* Concomitant chemotherapy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 296
Dates: Start 2001-03

PRIMARY OUTCOMES:
Late xerostomia rate

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Bardet, MD, Principal Investigator — Centre Régional de Lutte contre le Cancer de Nantes-Atlantique
Locations (1):
- Centre Régional de Lutte contre le Cancer de Nantes-Atlantique, Nantes, France

REFERENCES:
- [Background] Bardet E, Martin L, Calais G, Tuchais C, Bourhis J, Rhein B, Feham N, Alphonsi M. Preliminary data of the GORTEC 2000-02 phase III trial comparing intravenous and subcutaneous administration of amifostine for head and neck tumors treated by external radiotherapy. Semin Oncol. 2002 Dec;29(6 Suppl 19):57-60. doi: 10.1053/sonc.2002.37348. PMID 12577246